CLINICAL TRIAL: NCT05047588
Title: Stable Isotope Biomarker for Added Sugar Intake and Sweet Taste Phenotypes in Mother-child Dyads
Brief Title: Added Sugar Intake, Sweet Taste Phenotypes and Biomarkers
Acronym: SWBIO
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Responsible Party: Sponsor
Other Study IDs: 833299
Record Dates: First submitted 2021-08-13; First posted 2021-09-17 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: taste; children; dietary intake; biomarker; adult; sugar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of this cross-sectional study on a racially diverse group of children (3-10y) and their mothers are to determine whether the relationship between sweet taste phenotypes differed among mother-daughter and mother-son dyads and to determine the predictive value of a hair biomarker (delta13C). Given the widespread overconsumption of added sugars, and the associated burden of disease, improving surveillance measures and developing strategies to reduce added sugar intake, especially among the youngest members of society, are public health priorities.

DETAILED DESCRIPTION:
This is a single-site cross-sectional study designed to investigate the relationship of sweet taste phenotypes among mother-child dyads and assess the predictive value of a hair biomarker for sweet taste phenotypes. For each participant, we will collect 2-day 24-hour dietary recalls to determine added sugar intake; directly assess the level of sweet taste most preferred; measure liking/disliking of sweet tasting foods and beverages; collect anthropometric measures; and collect at least 3 cm of hair for biomarker analyses. Mothers will also complete a variety of questionnaires on parenting and child behavior.

ELIGIBILITY:
Inclusion Criteria:

* Hair that is greater than or equal to 3 cm in length
* Child is between the ages of 3 and 10 years and adult is between the ages of 18 and 70
* Access to electronic device including Smartphone, iPad, tablet, laptop, or desktop computer for participation in remote study visits.

Exclusion Criteria:

* Diagnosis of Type 2 Diabetes

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy adults and children
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Sweet taste preferences | Through study completion, average 2 and a half years
  Level of sucrose most preferred as determined by the Monell forced-choice tracking method [range of sucrose solutions: 0.09 to 1.05 M]
Diet intake | Through study completion, average 2 and a half years
  Two days of dietary intake will be obtained by having mothers report all the foods and beverage eaten during past day using the Automated Self-Administered Recall System (ASA24). Mothers will complete for herself and her child on two separate days. From these data, we will obtain daily energy intake (kcal/d), sugar (g/d; kcal/d) intake
PALS/ALS Liking surveys | Through study completion, average 2 and a half years
  Liking of different types of foods will by assessed by Preschool Adapted Liking Survey (PALS) for children [range -100 (maximal dislike) to 100 (maximal like)] and the Adult Liking Survey (ALS) for adults [range -100 (maximal dislike) to 100 (maximal like)]
Hair Biomarker for added sugar intake | After study completion, 2022
  Three cm of each hair sample will undergo stable isotope ratio mass spectrometry that will yield the concentration of carbon-13 relative to carbon-12 (added sugar biomarker, which has been shown to be associated with added sugar intake in older children and adults. Each cm reflects the added sugar intake of one month.

SECONDARY OUTCOMES:
Anthropometry | Through study completion, average 2 and a half years
  We will measure each participant's height (in cm) and weight (in kg). From these two measures, we will combine to calculate BMI (kg/m2) as well as determine the corresponding BMI-for-age percentile in children and BMI in adults.
Eating Behavior constructs | Through study completion, average 2 and a half years
  Mothers will complete the 35-item Adult Eating Behavior Questionnaire to describe her eating behaviors and the 26-item Children's Eating Behavior Questionnaire to describe her child's eating behaviors. Each item is scored from 1 (disagree/never) to 5 (agree/always) and are averaged and categorized into the following eating behavior constructs: enjoyment of food, food responsiveness, satiety responsiveness, emotional overeating; emotional undereating, and food fussiness. Higher numbers reflect more of the behavior.
Waist-to-Hip ratio | Through study completion, average 2 and a half years
  We will measure each participant's waist and hip in cm from which the ratio is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, PhD, Study Director — Monell Chemical Senses Center; Alissa D Smethers, RD PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Smethers AD, Fisher JO, Carney EM, Coffman DL, Mennella JA. Carbon stable isotope values in hair are associated with added sugar intake in adults but not young children: a cross-sectional study. Am J Clin Nutr. 2025 Apr;121(4):900-909. doi: 10.1016/j.ajcnut.2025.02.013. Epub 2025 Feb 18. PMID 39978470